CLINICAL TRIAL: NCT02009280
Title: A Comparison of Propofol Based Total Intravenous Anesthesia and Sevoflurane Based Balanced Anesthesia on Renal Protection During Lung Transplantation Under Extracorporeal Membrane Oxygenation - A Prospective, Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2013-0648
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Patients Undergoing Lung Transplantation Under Extracorporeal Membrane Oxygenation
Keywords: Propofol; Lung transplantation; Extracorporeal membrane oxygenation; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol group (Experimental): Propofol group
  Interventions: Drug: Administration of anesthesia: Propofol
- Sevoflurane group (Active Comparator): Sevoflurane group
  Interventions: Drug: Administration of anesthesia: Sevoflurane

INTERVENTIONS:
Drug: Administration of anesthesia: Propofol — Maintenance of anesthesia with the propofol
  Arms: Propofol group
Drug: Administration of anesthesia: Sevoflurane — Maintenance of anesthesia with the sevoflurane
  Arms: Sevoflurane group

SUMMARY:
The aim of this study is to investigate whether propofol based total intravenous anesthesia reduces incidence of acute kidney injury following the lung transplantation under extracorporeal membrane oxygenation

ELIGIBILITY:
Inclusion Criteria:

* Sixty adults undergoing lung transplantation under extracorporeal membrane oxygenation

Exclusion Criteria:

* Patient having propofol allergy, BMI > 30 kg/m2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the incidence of acute kidney injury between the lung transplantation recipients under propofol based anesthesia and inhalation based anesthesia | Postoperative 48 hours
  Developement of the acute kidney injury is determined by Plasma neutrophil gelatinase-associated lipocalin (NGAL), Cystatin C, and Creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea